CLINICAL TRIAL: NCT02940457
Title: Verbesserung Kognitiver Fähigkeiten Bei Personen Mit Verdacht Auf Eine Leichte Kognitive Beeinträchtigung
Brief Title: Cognitive Ability Training for Seniors With Mild Cognitive Impairment
Acronym: MICE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The employe for the study quit and a new grant proposal was not financed
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wuerzburg165/16
Record Dates: First submitted 2016-10-11; First posted 2016-10-21 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2019-04

CONDITIONS: Mild Cognitive Impairment
Keywords: tDCS; MCI; Working Memory; fNIRS
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum tDCS (Experimental): prefrontal anodal stimulation
  Interventions: Device: Verum tDCS
- Sham tDCS (Experimental): sham stimulation, same electrode positions
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Verum tDCS — Neuropsychological (working memory) training for 30 minutes, 6 sessions tDCS during training with 2 mA
  Arms: Verum tDCS
Device: Sham tDCS — Neuropsychological (working memory) training for 30 minutes, 6 sessions tDCS during training with 0 mA
  Arms: Sham tDCS

SUMMARY:
This study investigates the beneficial effects of prefrontal brain stimulation (with transcranial direct current stimulation [tDCS]) during working memory training in seniors with mild cognitive impairments.The placebo-controlled double blinded study includes 50 elderly patients which will be randomized into verum or sham tDCS.

DETAILED DESCRIPTION:
In this project, we want to test whether the effectiveness of neuropsychological exercise therapy can be increased in elderly persons suspected of having an MCI by means of parallel tDCS treatment.

All test participants train over 6 sessions within 2 weeks two different working memory tasks with increasing difficulty. In the randomized, double-blind, prospective therapy study, participants are assigned to either a Verum-tDCS or a placebo-tDCS group. The Verum-tDCS group receives active stimulation in parallel to the exercise therapy, while the placebo group does not receive tDCS stimulation. To check the effects of the therapy, we measure performance and neuronal activation in different executive tasks using near-infrared spectroscopy (NIRS). Furthermore, we will check whether the training increases the volume of the grey matter (Draganski et al., 2004, Malchow et al., 2016) and the expression of BDNF can be increased (Schuch et al., 2015).

ELIGIBILITY:
Inclusion Criteria:

* suspected MCI
* total CERAD score <= 85.1
* MMSE >=24
* native german speaker
* between 50-75 years old
* right handed

Exclusion Criteria:

* impairment of daily living activities
* psychiatric, neurological diseases
* uncorrected hearing or vision deficits
* actual psychopharmaca intake
* metal parts in the head
* medical electronical implants

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Brain activation measured with NIRS | 4 weeks
  The Investigators are measuring brain activation during executive functions
Reaction times, errors and number of generated words in neuropsychological tasks | 4 weeks
  The Investigators are measuring cognitive performance for different executive functions

SECONDARY OUTCOMES:
T1 weighted magnetic resonance Imaging (MRI) of the brain | 4 weeks
  Structural changes in grey matter of the brain calculated by voxel based morphometry (VBM)
Blood sampling | 4 weeks
  Increased BDNF secretion in serum

CONTACTS AND LOCATIONS:
Overall Officials: Martin Herrmann, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- University Hospital, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No